CLINICAL TRIAL: NCT05394519
Title: Efficacy and Safety of Cagrilintide s.c. 2.4 mg in Combination With Semaglutide s.c. 2.4 mg (CagriSema s.c. 2.4 mg/2.4 mg) Once-weekly in Participants With Overweight or Obesity and Type 2 Diabetes
Brief Title: A Research Study to See How Well CagriSema Helps People With Type 2 Diabetes and Excess Body Weight Lose Weight
Acronym: REDEFINE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4609; U1111-1267-4287 (Other: World Health Organization (WHO)); 2021-005121-24 (EudraCT Number); jRCT2031220671 (Registry Identifier: jRCT (Japan))
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CagriSema (Experimental): Cagrilintide + semaglutide once weekly
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Placebo (Placebo Comparator): Placebo cagrilintide + semaglutide once weekly
  Interventions: Drug: Placebo cagrilintide; Drug: Placebo semaglutide

INTERVENTIONS:
Drug: Cagrilintide — Cagrilintide administered subcutaneously (s.c., under the skin) once-weekly
  Arms: CagriSema
Drug: Semaglutide — Semaglutide administered subcutaneously (s.c., under the skin) once-weekly
  Arms: CagriSema
Drug: Placebo cagrilintide — Placebo cagrilintide administered subcutaneously (s.c., under the skin) once-weekly
  Arms: Placebo
Drug: Placebo semaglutide — Placebo semaglutide administered subcutaneously (s.c., under the skin) once-weekly
  Arms: Placebo

SUMMARY:
This study will look at how well the new medicine CagriSema helps people living with excess body weight and type 2 diabetes losing weight. Participants will either get CagriSema or a dummy medicine. Which treatment they get is decided by chance.

The study will last for about 1½ years. Women cannot take part if pregnant, breast-feeding or planning to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age above or equal to 18 years at the time of signing informed consent
* BMI greather than or equal to 27.0 kg/m^2
* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days before screening
* Treatment with either lifestyle intervention, or treatment with 1-3 marketed oral antidiabetic drugs (OAD)s (metformin, α-glucosidase inhibitors (AGI), glinides, sodium-glucose co-transporter 2 inhibitor (SGLT2i), thiazolidinediones, or sulphonylureas (SU)s as a single agent or in combination) according to local label
* Treatment with oral antidiabetic drugs should be stable (same drug(s), dose and dosing frequency) for at least 90 days before screening
* HbA1c 7%-10% (53-86 mmol/mol) (both inclusive) as measured by the central laboratory at screening

Exclusion Criteria:

* Clinically significant or severe hypoglycaemia within 6 months before screening or history of hypoglycaemia unawareness
* Renal impairment with estimated glomerular filtration rate (eGFR) below 30 mL/min/1.73 m^2, as measured by the central laboratory at screening
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%).
Achievement of greater than or equal to (≥) 5% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Count of participant.

SECONDARY OUTCOMES:
Achievement of ≥ 20% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Count of participant.
Relative change in body weight | From baseline (week 0) to week 20
  Measured in %.
Change in waist circumference | From baseline (week 0) to end of treatment (week 68)
  Measured in centimeter (cm).
Change in Glycated Haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 68)
  Measured in %-points.
Change in Systolic Blood Pressure (SBP) | From baseline (week 0) to end of treatment (week 68)
  Measured in millimeter of mercury (mmHg).
Change in Impact of Weight on Quality Of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function score | From baseline (week 0) to end of treatment (week 68)
  Measured in score points.
Change in Short Form-36 Version 2.0 Health Survey Acute (SF-36v2 Acute) Physical Functioning score | From baseline (week 0) to end of treatment (week 68)
  Measured in score points.
Change in body weight | From baseline (week 0) to end of treatment (week 68)
  Measured in kilogram (kg).
Change in body mass index (BMI) | From baseline (week 0) to end of treatment (week 68)
  Measured in kilogram per meter square (kg/m^2).
Improvement in weight category (BMI, underweight below 18.5, normal weight 18.5 to below 25, overweight 25.0 to below 30, obesity class I 30 to below 35, obesity class II 35 to below 40, obesity class III above 40) | From baseline (week 0) to end of treatment (week 68)
  Count of participant.
Achievement of HbA1c less than or equal to (≤) 6.5% | At end of treatment (week 68)
  Count of participant.
Change in Fasting Plasma Glucose (mmol/L) | From baseline (week 0) to end of treatment (week 68)
  Measured in millimoles per liter (mmol/L).
Change in Fasting Plasma Glucose (mg/dL) | From baseline (week 0) to end of treatment (week 68)
  Measured in milligram per deciliter (mg/dL)
Ratio to baseline in fasting serum insulin | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Change in Diastolic Blood Pressure (DBP) | From baseline (week 0) to end of treatment (week 68)
  Measured in mmHg.
Ratio to baseline in C-reactive protein (CRP) | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: Total cholesterol, High-density lipoprotein (HDL) cholesterol, Low-density lipoprotein (LDL) cholesterol, Very low-density lipoprotein (VLDL) cholesterol, Triglycerides and Free fatty acids | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Change in IWQOL-Lite-CT: Total score, Physical and Psycosocial score | From baseline (week 0) to end of treatment (week 68)
  IWQOL-Lite-CT is a 20-item clinical outcomes assessment (COA) instrument used to assess the impact of body weight changes in obesity studies on patients' physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score. Score ranges for composite score (physical composite, psychosocial composite and physical function composite) and Total score is 0-100. Higher scores indicate better level of functioning.
Change in Control of Eating Questionnaire (CoEQ): Craving Control score, Positive Mood score, Craving for Sweet score, Craving for Savoury food score, Hunger score and Satiety score | From baseline (week 0) to end of treatment (week 68)
  CoEQ is a 19-item multidimensional patient-reported outcome (PRO) that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), and craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). Higher score represents a greater level of Craving Control.
Achievement of at least 14.6-point increase (yes/no) in IWQOL-Lite-CT Physical Function score | From baseline (week 0) to end of treatment (week 68)
  Count of participant.
Achievement of at least 3.7-point increase (yes/no) in SF-36v2 Acute Physical Functioning score | From baseline (week 0) to end of treatment (week 68)
  Count of participant.
Change in IWQOL-Lite-CT Physical Function score | From baseline (week 0) to end of treatment (week 68)
Achievement of at least 14.6-point increase (yes/no) in IWQOL-Lite -CT Physical Function score for subgroup | From baseline (week 0) to end of treatment (week 68)
  Count of participant.
Continuous glucose monitoring: Change in mean glucose (mmol/L) | From baseline (week 0) to end of treatment (week 68)
  Measured in mmol/L.
Continuous glucose monitoring: Change in mean glucose (mg/L) | From baseline (week 0) to end of treatment (week 68)
  Measured in mg/L.
CGM: Change in time above range (TAR) >10.0 mmol/L (>180 mg/dL) | From baseline (week 0) to end of treatment (week 68)
  Measured in %-points.
CGM: Change in time in range (TIR) 3.9-10.0 mmol/L (70-180 mg/dL) | From baseline (week 0) to end of treatment (week 68)
  Measured in %-points.
CGM: Change in time above high range (TAHR) >13.9 mmol/L (>250 mg/dL) | From baseline (week 0) to end of treatment (week 68)
  Measured in %-points.
CGM: Change in time in tight range (TITR) 3.9-7.8 mmol/L (71-140 mg/dL) | From baseline (week 0) to end of treatment (week 68)
  Measured in %-points.
CGM: Within-day glycaemic variability (% CV) | At end of treatment (week 68)
  Measured in %.
Number of Treatment Emergent Adverse Events (TEAEs) | From baseline (week 0) to end of study (week 75)
  Count of events.
Number of Treatment Emergent Serious adverse events (TESAEs) | From baseline (week 0) to end of study (week 75)
  Count of events.
Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) | From baseline (week 0) to end of study (week 75)
  Count of episodes.
Number of severe hypoglycaemic episodes (level 3): hypoglycaemia associated with severe cognitive impairment requiring external assistance for recovery, with no specific glucose threshold | From baseline (week 0) to end of study (week 75)
  Count of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (177):
- United States (48):
  - John Muir Physicians Network, Concord, California
  - Headlands Research California, LLC, Escondido, California
  - Providence Medical Foundation, Fullerton, California
  - St. Jos Heritage Hlthcr_Fllrtn, Fullerton, California
  - Diabetes/Lipid Mgmt & Res Ctr, Huntington Beach, California
  - Clinical Trials Research, Lincoln, California
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - Velocity Clin Res Wstlke, Los Angeles, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - New West Physicians,Inc., Golden, Colorado
  - Clinical Res Of W Florida Inc, Clearwater, Florida
  - Northeast Research Institute, Fleming Island, Florida
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - Renstar Medical Research, Ocala, Florida
  - AdventHealth Diab Inst, Orlando, Florida
  - Florida Institute for Clinical Research, LLC, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Endo Res Solutions Inc, Roswell, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - Cotton-Oneill Diabetes and End, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Pennington Biom Res Ctr, Baton Rouge, Louisiana
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Mercury Str Med Grp, PLLC, Butte, Montana
  - AMC Community Endocrinology, Albany, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Texas Diab & Endo, P.A., Austin, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - National Clin Res Inc., Richmond, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Amherst Family Practice P.C., Winchester, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington
- Austria (6):
  - Universitätsklinik für Innere Medizin Graz, Graz
  - Barmh. Brüder Linz, Konventspital, Linz
  - Fließer-Görzer [Ordination], Saint Stefan
  - Klinik Landstraße, Vienna
  - Universitätsklinikum AKH Wien, Vienna
  - Imed 19- privat, Vienna
- Canada (13):
  - LMC Clin Res Inc. Calgary, Calgary, Alberta
  - C-endo Diab Endo Clin Calgery, Calgary, Alberta
  - Dr. M.B. Jones Inc, Victoria, British Columbia
  - Commonwealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - Dr. Harpreet Bajaj, Brampton, Ontario
  - Centricity Research Etobicoke Endocrinology, Etobicoke, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Milestone Research, London, Ontario
  - LMC Research Inc. Ottawa, Nepean, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Centre Medical Acadie, Montreal, Quebec
  - Centricity Res Pointe-Claire, Pointe-Claire, Quebec
  - LMC Clin Rsrch Inc. (Montreal), Saint-Laurent, Quebec
- Germany (10):
  - Diabetespraxis Mergentheim, Bad Mergentheim
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung GmbH, Essen
  - Universitätsklinikum Freiburg - Innere Medizin II, Freiburg im Breisgau
  - Wendisch - Dahl Hamburg - DZHW, Hamburg
  - AmBeNet GmbH, Leipzig
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
  - MZM Praxis Drs. Erlinger, Stuttgart
  - Zentrum für klinische Studien Allgäu Oberschwaben, Wangen
- Hungary (9):
  - Szegedi Tudomanyegyetem St Györgyi Albert Klinikai Központ, Szeged, Csongrád-Csanád
  - Debreceni Egyetem Belgyógyászati Klinika, Debrecen, Hajdú-Bihar
  - Hetényi Géza Kórház, Szolnok, Jász-Nagykun-Szolnok
  - Komáromi Selye János Kórház, Komárom, Komárom-Esztergom
  - Clinexpert Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - Szőcs Depot Egészségügyi Szolgáltató Kft., Budapest
  - Bajcsy-Zsilinszky Kórház, Budapest
  - Selye János Kórház és Rendelőintézet, Komárom
  - Hetényi Géza Kórház, Szolnok
- India (20):
  - HCG Hospitals, Ahmedabad, Gujarat
  - Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Calicut Medical College, Kozhikode, Kerala
  - Indian Institute of Diabetes, Thiruvnanthapuram, Kerala
  - Excel Endocrine Centre, Kolhāpur, Maharashtra
  - BYL Nair Hospital and T N Medical College Department of endo, Mumbai, Maharashtra
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Sunil's Diabetes Care n' Research Centre Pvt Ltd, Nagpur, Maharashtra
  - Noble Hospitals Pvt Ltd., Pune, Maharashtra
  - All India Institute of Medical Sciences_Delhi, Ansārinagar, New Delhi
  - Post Graduate Institute of Medical Education & Research_Chandigarh, Chandigarh, Punjab
  - J K Lon Hospital, SMS Medical College & Attached Hospitals, Jaipur, Rajasthan
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Apollo Research & Innovation (ARI), Chennai, Tamil Nadu
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Gleneagles Hospitals, Hyderabad, Telangana
  - Apollo Multispeciality Hospital, Kolkata, Kolkata, West Bengal
  - Apollo Multispeciality Hospitals Limited, Kolkata, West Bengal
  - Sunil's Diabetes Care n' Research Centre Pvt Ltd, Nagpur
  - Lady Hardinge Medical College, New Delhi
- Ireland (7):
  - CRF - Galway, Galway, Connaght
  - CRF HRB - Galway, Galway, Connaght
  - Clinical Research Centre, St. Vincent's University Hospital,, Dublin, Leinster
  - Mater Miscericordiae Hospital, Dublin, Leinster
  - St James's CRF, Dublin, Leinster
  - Connolly Hospital_Blanchardstown_Diabetes Day Centre, Dublin, Leinster
  - Connolly Hospital, Dublin, Leinster
- Japan (6):
  - TOSAKI Clinic for Diabetes and Endocrinology_Diabetes and Endocrinology, Aichi
  - Tokuyama clinic_Diabetic internal medicine, Chiba
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Osaka Nishiumeda Clinic_Diabetes Internal Medicine, Osaka
  - Osaka University Hospital_Metabolic Medicine, Osaka
  - Takatsuki Red Cross Hospital, Osaka
- Malaysia (10):
  - Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan
  - Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur
  - Hospital Seri Manjung, Seri Manjung, Perak
  - Hospital Putrajaya, Putrajaya, Putrajaya
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Miri, Miri, Sarawak
  - Hospital Ampang, Ampang, Selangor, Selangor
  - University Technology MARA (UiTM) - Sg Buloh, Sungai Buloh, Selangor
  - Hospital Melaka, Malacca
  - Hospital Tuanku Jaafar, Seremban
- Poland (20):
  - Gierach-Med, Bygdoszcz, Kuyavian-Pomeranian Voivodeship
  - Linden sp. z o.o. sp. k., Krakow, Lesser Poland Voivodeship
  - Beata Miklaszewicz & Dariusz Dabrowski "CARDIAMED" s.j., Legnica, Lower Silesian Voivodeship
  - Terpa Sp. z o.o. Sp. k., Lublin, Lubelskie Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Im. Prof. W. Orłowskiego Centrum Medycznego Kształcenia Podyplomowego, Warsaw, Masovian Voivodeship
  - Medical Concierge Centrum Medyczne, Warsaw, Masovian Voivodeship
  - Instytut Diabetologii Sp. z o.o., Warsaw, Mazovian Voivodeship
  - Instytut Diabetologii Sp. z o.o., Warsaw, Mazovian
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Gabinet Leczenia Otylosci i Chorob Dietozaleznych, Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Salvia, Katowice, Slaskie Voivodeship
  - Klinika Bellamed, Elblag, Warmian-Masurian Voivodeship
  - Centrum Zdrowia Metabolicznego, Poznan, Wielkopolskie Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Gierach-Med, Bygdoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Linden sp. z o.o. sp. k., Krakow
  - Terpa Sp. z o.o. Sp. k., Lublin
  - Trialmed CRS, Piotrkow Trybunalski, Łódź Voivodeship
- Ponce Med School Found Inc, Ponce, Puerto Rico
- Thailand (10):
  - Siriraj Hospital_Bangkoknoi, Bangkok, Bangkoknoi, Bangkok, Bangkok
  - Ramathibodi Hospital, Bangkok, Ratchathewi Bangkok
  - King Chulalongkorn Memorial Hospital_Bangkok, Bangkok
  - King Chulalongkorn Memorial Hospital_Endocrinology, Bangkok
  - Rajavithi Hospital_Diabetes and Endocrinology, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital_Dept Endocrinology, Bangkok
  - Srinagarind Hospital, Khon Kaen
  - Thammasat Hospital_Cardiology, Pathum Thani
- United Kingdom (17):
  - Harrogate District Hospital, Harrogate, North Yorkshire
  - Crouch Oak Family Practice, Addlestone, Surrey
  - Antrim Area Hospital, Antrim
  - Layton Medical Centre, Blackpool
  - The Health Centre, Bradford-on-Avon
  - Southmead Hospital, Bristol
  - Hathaway Medical Centre, Chippenham
  - HMC Health - Heston, Hounslow
  - Leicester General Hospital, Leicester
  - Kiltearn Medical Centre, Nantwich
  - Clifton Medical Centre, Rotherham
  - Ashfields Primary Care Centre, Sandbach
  - Staploe Medical Centre, Soham
  - Joint Clinical Research Facility - Swansea, Swansea
  - Musgrove Park Hospital, Taunton
  - Royal Cornwall Hospital (Treliske), Truro
  - Albany House Medical Centre, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Davies MJ, Bajaj HS, Broholm C, Eliasen A, Garvey WT, le Roux CW, Lingvay I, Lyndgaard CB, Rosenstock J, Pedersen SD; REDEFINE 2 Study Group. Cagrilintide-Semaglutide in Adults with Overweight or Obesity and Type 2 Diabetes. N Engl J Med. 2025 Aug 14;393(7):648-659. doi: 10.1056/NEJMoa2502082. Epub 2025 Jun 22. PMID 40544432